CLINICAL TRIAL: NCT07093281
Title: The Impact of Live Attenuated Intranasal Influenza Vaccine Exposure on Mucosal Immunity
Brief Title: Intranasal LAIV Mucosal Immunity Examination
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Adam Kaufman, Assistant Professor of Otolaryngology, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HP-00114022
Record Dates: First submitted 2025-07-14; First posted 2025-07-30 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Impact of Vaccination
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional LAIV (Experimental): Intranasal Flu Vaccine
  Interventions: Biological: Live Attenuated Influenza Vaccine
- No Intervention (No Intervention): No Intervention

INTERVENTIONS:
Biological: Live Attenuated Influenza Vaccine — Nasal spray
  Arms: Interventional LAIV

SUMMARY:
The research of the investigators is focused on the understanding how the immune system functions and responds to intranasal vaccines. Intranasal vaccines do not lead to the same changes in the blood that intramuscular vaccines do. Therefore, the investigators want to look at the function of immune (lymphoid) organs that are near the nose. The closest immune organs are the adenoids and tonsils. Mice do not have tonsils allowing for the investigators to answer these questions. Human lymphoid tissue will allow the investigators to better understand the molecular behavior of these cells in humans.

The purpose of this protocol is to administer the FDA approved live attenuated influenza vaccine or no vaccine to patients undergoing adenoidectomy and/or tonsillectomy for obstructive sleep apnea prior to surgery and then collect the tissue (adenoid and/or tonsil tissue) that would normally be discarded from surgery. This will allow for improved understanding of what happens after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing tonsillectomy and adenoidectomy as part of the standard of care for sleep apnea

Exclusion Criteria:

* Chronic Tonsillitis
* Immune Deficiency
* Already received this year's flu vaccine

Ages: 2 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Serological outcomes will be compared before and after vaccination and between groups. | From enrollment to 4 weeks after surgery is completed
  The comparisons will specifically compare:
  Mean HAI Ab titers in serum and mucosal secretions

SECONDARY OUTCOMES:
Hemagglutinin Levels | From enrollment to 4 weeks after surgery
  Mean HA IgG and IgA titers in serum and mucosal secretions
Neuraminidase Levels | From enrollment to 4 weeks after surgery
  Mean NA IgG and IgA titers in serum and in mucosal secretions
Influenza Specific Antibodies | From enrollment to 4 weeks after surgery
  Non-neutralizing influenza-specific antibody titers before and after vaccination
Seroconversion rats | From enrollment to 4 weeks post surgery
  Comparison of serconversion rates

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States